CLINICAL TRIAL: NCT06978283
Title: The Effect of Artificial Intelligence-assisted Visual Case Analysis on Nursing Students' Knowledge and Attitudes Towards Pressure Injury Prevention: A Single-blind Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Çankırı Karatekin University (Other)
Responsible Party: Principal Investigator, Gözde ÖZARAS ÖZ, Principal Investigator, Çankırı Karatekin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: E-52950036-199-238039
Record Dates: First submitted 2025-05-03; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Artificial Intelligence (AI); Visual Case Analysis; Nursing Students; Pressure Injury Prevention; A Single-blind Randomized Controlled Trial
Keywords: AI-assisted; visual case analysis; Nursing Students; Artificial Intelligence (AI); pressure injury prevention; randomized controlled trial

STUDY DESIGN:
Intervention Model Description: This study will conduct as a single-blind randomized controlled trial according to the CONSORT guideline to evaluate the effect of AI-assisted visual case analysis on nursing students' knowledge and attitudes towards pressure injury prevention.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Artificial intelligence (Experimental): Nursing students will be provided with pressure injury prevention training using AI-assisted visual case analysis. The cases will be analyzed through an AI-assisted platform, and the students' knowledge and attitude levels were assessed.
  Interventions: Behavioral: AI-assisted case analysis
- Traditional case analysis (Active Comparator): Pressure injury prevention training will be given to nursing students using the traditional case analysis method. Case analysis will be performed using written materials.
  Interventions: Behavioral: Traditional case analysis

INTERVENTIONS:
Behavioral: AI-assisted case analysis — Nursing students will perform visual case analyses of pressure injuries using an AI-based platform. The AI system will provide students with case-based feedback.
  Arms: Artificial intelligence
Behavioral: Traditional case analysis — Participants will be present with written case scenarios and a case analysis will conduct with the instructor. The training process will be carried out with group discussions and the instructor's guidance. No technological or artificial intelligence support will be used.
  Arms: Traditional case analysis

SUMMARY:
The goal of this clinical trial is to examine the effect of artificial intelligence-assisted visual case analysis on nursing students' knowledge and attitudes towards pressure injury prevention. The main hypotheses it aims to answer are:

* AI-assisted visual case analysis affects nursing students' knowledge about pressure injury prevention.
* AI-assisted visual case analysis affects nursing students' attitudes toward pressure injury prevention.

Researchers will compare AI-assisted case analysis to conventional case analysis to see if it affected nursing students' knowledge and attitudes about pressure injury prevention.

Participants,

* The case group will shown an AI-supported presentation explaining the pressure injury prevention case. The control group will given a classic case analysis.
* At the end of the case, the PUPKAI and APuP scales will administered to the students in written form in the classroom.

ELIGIBILITY:
Inclusion Criteria:

* Taking the Fundamentals of Nursing II course for the first time
* Not working as a nurse in a health institution.
* Volunteering to participate in the study.

Exclusion Criteria:

* Having previously received patient pressure injury prevention training;
* Having repeated the Fundamentals of Nursing II course;
* Having difficulty speaking and understanding Turkish;
* Exceeding the course attendance time
* Not attending pressure injury prevention training and evaluation
* Filling in incomplete data
* Graduating from a health-related high school or university.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-05-09 (Estimated); Primary Completion 2025-05-09 (Estimated); Study Completion 2025-07-10 (Estimated)

PRIMARY OUTCOMES:
The Pressure Ulcer Prevention Knowledge Assessment Instrument (PUPKAI) | Day 1
  The PUPKAI was developed by Beeckman and colleagues. It includes six subscales: etiology and development, classification and monitoring, risk assessment, nutrition, preventive interventions to reduce the amount of pressure/slip, and preventive measures to reduce the duration of pressure/slip. Each question has three answer options, one of which is correct. The total number of correct answers for each subscale and the entire instrument indicates the level of knowledge. The maximum score that can be obtained from the instrument is 26, and the acceptable score for proficiency is ≥ 16 (60%). The validity and reliability of the instrument in the Turkish population was tested by Tulek and colleagues. The content validity index of the instrument was 0.94. The internal consistency reliability for the overall instrument was determined using the Kuder-Richardson test. The Kuder-Richardson-20 value was 0.80.

SECONDARY OUTCOMES:
Attitude Towards Pressure Ulcer Prevention Device (APuP) | Day 1
  APuP was developed by Beeckman and colleagues from Ghent University in Belgium in 2010 to examine the attitudes of nursing students towards the prevention of pressure injuries. The scale consists of five sub-dimensions and 13 items. The sub-dimensions are "attitude towards personal competence in preventing pressure injuries", "attitude towards the priority of preventing pressure injuries", "attitude towards the impact of pressure injuries", "attitude towards personal responsibility in preventing pressure injuries" and "attitude towards the effectiveness of prevention". Items 3, 5, 7, 8, 9, 10 and 13 are reverse scored. The scores on the scale range from 13 to 52. An average attitude score of more than 75% is considered satisfactory. High total APuP scores indicate positive attitudes. The validity and reliability study of the scale for the Turkish population was conducted by Üstün in 2013.

CONTACTS AND LOCATIONS:
Locations (1):
- Cankiri Karatekin University. Faculty of Health Sciences., Çankırı, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Due to participant privacy protection and ethics committee restrictions, IPD sharing is not planned.